CLINICAL TRIAL: NCT04293978
Title: Virtual Reality Relaxation at an Adolescent Addiction Inpatient Ward: A Single-arm Pilot Trial
Brief Title: Virtual Reality Relaxation for Addiction Inpatients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment and intervention provision paused due to COVID-19 situation. Planned to resume.
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm University (Other)
Responsible Party: Principal Investigator, Philip Lindner, Head of Research and Development, Maria Ungdom Clinic, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Virtuella Lugna rummet
Record Dates: First submitted 2020-02-21; First posted 2020-03-03 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Addiction
Keywords: Virtual Reality; Relaxation
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Single-arm, with immediate effects of interest. Varying number of intervention uses across participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality relaxation (Experimental): Participants may request to use the application at any time during their stay at the ward, as many times as they wish. Participants sign in using an anonymous study ID and sessions (and outcomes) are automatically logged by the device to this ID.
  Interventions: Behavioral: CalmPlace

INTERVENTIONS:
Behavioral: CalmPlace — Self-contained VR application allowing the user to build and custom a relaxation session, with options to vary session length (9-20 minutes), music/sound, relaxation exercises, and specific nature environment (three available) including time of day and events (e.g. rain). Delivered using an Oculus Go devices in kiosk-mode.

SUMMARY:
This trial examines the immediate session effect of Virtual Reality (VR) relaxation, when used at an addiction inpatient ward for adolescents.

DETAILED DESCRIPTION:
Past research has revealed that Virtual Reality nature environments can be used to induce relaxation, yet this type of intervention has not yet been evaluated in a clinical setting. This trial examines whether VR relaxation can be used as a digital equivalent of a (physical) comfort room at an an addiction inpatient ward for adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Maria Ungdom inpatient ward.
* Sufficient grasp of Swedish to understand terms of study participation and intervention instructions.

Exclusion Criteria:

* Self-reported stereoscopic vision or balance problems hindering VR experience.
* Self-reported history of repeated violent outbursts when using technology.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in general well-being | Change from baseline (start of session) to immediately after the intervention
  Rated 0-100 using a visual analogue scale with smiley-type anchors (higher score is better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lindner, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Maria Ungdom Heldygnsvård, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Raw outcome data (with no other identifiable information) may be shared with other researchers under conditions described below.
Supporting Information: Analytic Code
Time Frame: When trial is published and up to ten years after that.
Access Criteria: Signed data sharing agreement.

REFERENCES:
- [Background] Lindner P, Miloff A, Hamilton W, Carlbring P. The Potential of Consumer-Targeted Virtual Reality Relaxation Applications: Descriptive Usage, Uptake and Application Performance Statistics for a First-Generation Application. Front Psychol. 2019 Feb 4;10:132. doi: 10.3389/fpsyg.2019.00132. eCollection 2019. PMID 30778311